CLINICAL TRIAL: NCT02734745
Title: Accuracy of Flash Glucose Monitoring Freestyle Libre (Abbott) in Home Setting and In-patient Setting During Hypo - Hyperglycemia
Brief Title: Accuracy of Freestyle Libre
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Daniela Bruttomesso, medical doctor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3724/AO/16
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Type 1
Keywords: diabetes type 1; flash glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- flash glucose monitoring (Experimental): Patients will use a device: Freestyle Libre for 14 days
  Interventions: Device: flash glucose monitoring

INTERVENTIONS:
Device: flash glucose monitoring — Patients will use Freestyle Libre for 14 days at home, during this period they will have to perform at least 7 measurements of capillary blood glucose per day . Patients also will go to our clinical center on two separate occasions , to run a test breakfast. In one of the two occasions it will be specifically induced a moderate initial hyperglycemia and subsequent hypoglycemia . During the test meal and in the subsequent hours for a total of 6 hours , will be carried out frequent blood sampling for measurement of blood glucose using the Yellow Springs glucose analyzer ( YSI system ) , simultaneous measurements with Freestyle Libre and with glucometer.

SUMMARY:
This is an open-label, mono-centre, interventional study.The aim of this trial is to assess accuracy and reliability of a flash glucose monitoring system, the freestyle Libre (Abbott, CA, USA), in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Objective: To assess accuracy and reliability of a new-to-market flash glucose monitoring system, the freestyle Libre (Abbott, CA, USA), in patients with type 1 diabetes.

Study design: open-label, mono-centre interventional study. Patients will wear freestyle Libre for 14 days in the home setting. There will be no limitations in food intake or in physical activity, but patients will have at least 7 finger-stick/days. Patients will have 2 visits in our clinical center and in these visits we'll compare freestyle Libre values with blood sampling to determine glucose values with YSI, during euglycemia and during glucose excursion and induced hypo-hyperglycemia.

Study population: 48 patients will be included in this trial. Every patient will wear device for 14 days at home and during 2 visits at CRC Study endpoints: main endpoint will be the evaluation of freestyle Libre accuracy during real life compared to glucometer values and to YSI glucose values (during 2 visits). A separate analysis will be performed on the accuracy of the freestyle Libre in the hypoglycaemic (defined as a blood glucose value ≤3.9 mmol/L) and hyperglycaemic area (defined as a blood glucose value ≥10.0 mmol/L). Additionally, a separate analysis will be performed to assess device performance and accuracy per day of device life.

If patients enrolled in the study use Dexcom G4 or G5 (CGM) and wanted to continue to use it, he/she can do so. In this case we can compare the accuracy of Libre even towards Dexcom G4/G5 device.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of diabetes mellitus type 1 ( diagnosed according to World Health Organization criteria ) for at least one year
* Body Mass Index ( BMI ) < 35 kg / m²
* Willingness to wear the device and to comply with the study protocol during the entire duration of the same
* No restrictions linked to glycated hemoglobin ( HbA1c )
* Signature of informed consent before any study-related procedure

Exclusion Criteria:

* Pregnancy, breast-feeding, planning pregnancy, or refuse to use contraception during the study period (for female subjects).
* Known allergies to patches or skin disinfectants used during the study.
* skin lesions, irritation, redness, edema, in the possible application of the sensor sites that may interfere with the placement of the device or the detection accuracy of test results.
* blood donations in the 3 months preceding the study.
* Use of drugs that can interfere with glucose metabolism (such as steroids) unless it is chronic therapies whose dosage has remained stable over the last 3 months and is expected to remain stable during the study period.
* serious medical or psychological conditions that in the opinion of the medical team could compromise patient safety during study participation.
* Patients enrolled in other clinical trials.
* known disorders of the adrenal glands, pancreatic tumors, or insulinomas
* Inability of the patient to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of freestyle Libre flash monitoring | 14 days
  accuracy of freestyle Libre flash monitoring measured as MARD respect to blood glucose (YSI) during CRC visit and respect to glucometer during home setting

SECONDARY OUTCOMES:
Evaluate the accuracy of the Free Style Libre for each day of use and during normoglycaemia ( between 70 and 180 mg / dl ) | 14 days
  accuracy of freestyle Libre flash monitoring during normoglycaemia (between 70 and 180 mg / dl) measured as MARD respect to blood glucose (YSI) during CRC visit and respect to glocometer during home setting, accuracy for each day of use measured as MARD respect to glucometer
Evaluate the accuracy of the Free Style Libre for each day of use and during hypoglicaemia ( < 70 mg / dl ) | 14 days
  accuracy of freestyle Libre flash monitoring during hypogliacemia (< 70 mg / dl) measured as MARD respect to blood glucose (YSI) during CRC visit and respect to glucometer during home setting,
Evaluate the accuracy of the Free Style Libre for each day of use and during hyperglicemia ( >180 mg / dl ) | 14 days
  accuracy of freestyle Libre flash monitoring measured as MARD respect to blood glucose (YSI) during CRC visit and respect to glucometer during home setting,

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boscari F, Galasso S, Acciaroli G, Facchinetti A, Marescotti MC, Avogaro A, Bruttomesso D. Head-to-head comparison of the accuracy of Abbott FreeStyle Libre and Dexcom G5 mobile. Nutr Metab Cardiovasc Dis. 2018 Apr;28(4):425-427. doi: 10.1016/j.numecd.2018.01.003. Epub 2018 Jan 31. No abstract available. PMID 29502924
- [Derived] Fadini GP, Boscari F, Cappellari R, Galasso S, Rigato M, Bonora BM, D'Anna M, Bruttomesso D, Avogaro A. Effects of Hypoglycemia on Circulating Stem and Progenitor Cells in Diabetic Patients. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1048-1055. doi: 10.1210/jc.2017-02187. PMID 29300991
- [Derived] Boscari F, Galasso S, Facchinetti A, Marescotti MC, Vallone V, Amato AML, Avogaro A, Bruttomesso D. FreeStyle Libre and Dexcom G4 Platinum sensors: Accuracy comparisons during two weeks of home use and use during experimentally induced glucose excursions. Nutr Metab Cardiovasc Dis. 2018 Feb;28(2):180-186. doi: 10.1016/j.numecd.2017.10.023. Epub 2017 Nov 11. PMID 29258716